CLINICAL TRIAL: NCT00030355
Title: A Phase I/II Open-Label Study Of The Intravenous Administration Of Homoharringtonine (CGX-635) Salvage Therapy For The Treatment Of Refractory Acute Promyelocytic Leukemia
Brief Title: Homoharringtonine in Treating Patients With Refractory Acute Promyelocytic Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069158; CHEMGENEX-CGX-635-APL-101; MDA-DM-01265
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2007-09

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3); adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute | interventions — Homoharringtonine; Drug Therapy

INTERVENTIONS:
Drug: homoharringtonine
Procedure: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of homoharringtonine in treating patients who have refractory acute promyelocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of salvage therapy comprising homoharringtonine in patients with refractory acute promyelocytic leukemia.
* Determine the antileukemic efficacy of this drug in these patients.

OUTLINE: Patients receive remission induction therapy comprising homoharringtonine (HH) IV continuously on days 1-14. Courses repeat every 4 weeks in the absence of unacceptable toxicity until a complete remission (CR) is achieved or the patient fails to respond after 3 courses.

Patients who achieve a CR during induction therapy receive maintenance therapy comprising HH IV continuously on days 1-7. Maintenance treatment repeats every 4 weeks for a total of 12 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A maximum of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute promyelocytic leukemia confirmed morphologically and by t(15;17) translocation or molecular polymerase chain reaction
* Refractory to tretinoin, anthracyclines, and arsenic-based therapy (including arsenic trioxide) and for which no other alternative therapy of higher priority is appropriate

PATIENT CHARACTERISTICS:

Age:

* 12 and over

Performance status:

* Zubrod 0-3

Life expectancy:

* More than 4 weeks

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No active ischemia
* No other uncontrolled cardiac condition (e.g., angina pectoris, cardiac arrhythmia, hypertension, or congestive heart failure)
* No myocardial infarction within the past 12 weeks

Other:

* No other concurrent illness that would preclude study
* No other active malignancy
* No uncontrolled active infection
* No clinically significant screening serum chemistry results unless attributed to acute promyelocytic leukemia
* No medical or psychiatric condition that would preclude informed consent or study therapy
* HIV negative
* HTLV-I and HTLV-II negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior or concurrent leukapheresis allowed

Chemotherapy:

* See Disease Characteristics
* At least 15 days since prior systemic chemotherapy unless leukemia progression necessitates early therapy
* No other concurrent systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Recovered from prior therapy
* At least 15 days since other prior antileukemic therapy unless leukemia progression necessitates early therapy
* No other concurrent antileukemic therapy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety by physical examinations, vital signs, laboratory studies (routine hematology, clinical chemistry, pharmacokinetics, urinalysis, chest x-ray, and EKG), and solicited and unsolicited adverse events
Efficacy by response to treatment

SECONDARY OUTCOMES:
Pharmacokinetics
Duration of treatment response
Survival
Induction mortality
Hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States